CLINICAL TRIAL: NCT04634474
Title: The Effect of Closed System Suction on Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Zuhal Gülsoy, Dr, Cumhuriyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Zuhal Gülsoy
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Endotracheal Suction; Pain
Keywords: endotracheal suction, ,; pain,; behavioral pain scale
MeSH Terms: conditions — Pain | interventions — Suction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain on Endotracheal Suction (Experimental): Before and after endotracheal aspiration, the pain of the patient will be evaluated according to the DAS and VAS scale. VAS scores will be compared with DAÖ scores. Aspiration process will be applied to all patients by the same nurse. According to the DAQ, the pain will be assessed by a volunteer nurse who is not a researcher.
  Interventions: Behavioral: Suction

INTERVENTIONS:
Behavioral: Suction — Is DAS an accurate pain descriptor for every application in intensive care unit?;. This question guides the study. This study was planned with the thought that the result may be misleading in applications such as eye care and aspiration that will trigger reflex movements in intensive care. In addition, creating new evidence on whether endotracheal suction is a painful application is the basis of the application.

SUMMARY:
Endotracheal intubation and mechanical ventilation are life-saving practices in patients with respiratory failure, and aspiration of secretions is often required to maintain airway patency. Although tracheal aspiration is an unavoidable requirement to maintain airway patency, it can bring many undesirable conditions. In the presence of complications, the duration of hospital stay is also prolonged. In the literature, endotracheal aspiration is defined as a painful and uncomfortable method for patients. However, pain is an undesirable sensation that cannot be adapted. The most reliable source for pain assessment is the patient himself. However, verbal communication with patients in the ICU is quite difficult due to reasons such as the presence of endotracheal tube and tracheostomy, confusion, mechanical ventilation, and sedative drug use. Therefore, intensive care patients may not be able to express their pain verbally. In this case, patient behavior becomes important in pain assessment. Scales were developed for pain assessment of patients who could not express their pain. The "Behavioral Pain Scale" (DAS) was developed by Payen et al. For this purpose and made available to intensive care patients.

Patients who meet the inclusion criteria and agree to participate in the study when aspirating is required (Seeing pulmonary secretions in the endotracheal tube, tachypnea, tachycardia, hypertension, worsening of oxygen saturation and / or arterial blood gas, sawtooth pattern in the flow volume loop of the ventilator monitor and / or trachea Hearing of coarse breathing sounds, Ppeak inspiratory pressure increase in mechanical ventilator in volume-controlled mode, or tidal volume decrease in pressure-controlled mode, etc.) by a volunteer nurse, whether there is pain before, during and after aspiration, the severity and localization of the pain will be recorded by VAS and VAS. . The patient will be aspirated with the same aspiration technique in all patients by using a closed system aspiration catheter by the other volunteer nurse. Aspiration procedure will be applied to each patient according to the American association for respiratory care (AARC) aspiration guideline. The nurse evaluating the pain will record whether the patients have pain with DAS and VAS, the severity and localization of the pain

DETAILED DESCRIPTION:
Endotracheal intubation and mechanical ventilation are life-saving practices in patients with respiratory failure, and aspiration of secretions is often required to maintain airway patency. Although tracheal aspiration is an unavoidable requirement to maintain airway patency, it can bring many undesirable conditions. In the presence of complications, the duration of hospital stay is also prolonged. In the literature, endotracheal aspiration is defined as a painful and uncomfortable method for patients. However, pain is an undesirable sensation that cannot be adapted.

It is thought that performing aspiration in accordance with the AARC guideline and listening to music during the procedure reduce the pain in edotracheal aspiration. The most reliable source for pain assessment is the patient himself. However, verbal communication with patients in the ICU is quite difficult due to reasons such as the presence of endotracheal tube and tracheostomy, confusion, mechanical ventilation, and sedative drug use. Therefore, intensive care patients may not be able to express their pain verbally. In this case, patient behavior becomes important in pain assessment. Scales were developed for pain assessment of patients who could not express their pain. The "Behavioral Pain Scale" (DAS) was developed by Payen et al. For this purpose and made available to intensive care patients. DAS consists of three parts, including facial expression, upper extremity movements, and compliance with mechanical ventilation, and a total of 12 items. Each section is given a score between 1 and 4. The lowest pain score obtained from the scale is 3 and the highest pain score is 12. (Appendix 1) Patients with an unconscious communication can be established with a sign or writing method instead of verbal communication with patients with tracheostomy or tracheal tube. These patients can describe their pain without words. Visual pain scales can be used for this purpose. Visual Pain Scale (VAS) is one of these scales. VAS was first used in the 1970s. The scale was defined by Selby et al. To evaluate the quality of life in patients with cancer in the 1980s. VAS has been used in many studies evaluating different parameters after the 1990s and has recently been used in the measurement of special conditions such as pain. The test has proven itself for a long time and is a accepted test in the world literature. Safe, easy to apply Is DAS an accurate pain descriptor for every application in intensive care unit?;. This question guides the study. This study was planned with the thought that the result may be misleading in applications such as eye care and aspiration that will trigger reflex movements in intensive care.

6-Research protocol, materials and methods: METHOD In this study, when alpha 0.05, = 0.10, 1-B 0.90 was taken, 32 patients were included in the study and the power of the test was found to be P = 0.9657.

Time of Research: Research 01.07. It will be applied in the Anesthesia and Reanimation Intensive Care Unit (EIB) of a university hospital between 2020 - 31.12.2020.

The Type and Purpose of the Study: This study was planned as a prospective observational study in order to examine whether conscious patients connected to mechanical ventilator in the Anesthesia Intensive Care Unit experience pain during the closed system aspiration procedure, and if pain is experienced, whether NAC is reliable in evaluating the pain occurring in endotracheal aspiration.

The Population and Sample of the Study: The population of the study was the sample of all patients who were treated in the Anesthesia and Reanimation Intensive Care unit of a university hospital between the research dates, and the patients who were connected to the ventilator who agreed to participate in the study and underwent endotracheal aspiration.

Research Application Patients who meet the inclusion criteria and agree to participate in the study when aspirating is required (Seeing pulmonary secretions in the endotracheal tube, tachypnea, tachycardia, hypertension, worsening of oxygen saturation and / or arterial blood gas, sawtooth pattern in the flow volume loop of the ventilator monitor and / or trachea Hearing of coarse breathing sounds, Ppeak inspiratory pressure increase in mechanical ventilator in volume-controlled mode, or tidal volume decrease in pressure-controlled mode, etc.) by a volunteer nurse, whether there is pain before, during and after aspiration, the severity and localization of the pain will be recorded by VAS and VAS. . The patient will be aspirated with the same aspiration technique in all patients by using a closed system aspiration catheter by the other volunteer nurse. Aspiration procedure will be applied to each patient according to the American association for respiratory care (AARC) aspiration guideline. The nurse evaluating the pain will record whether the patients have pain with DAS and VAS, the severity and localization of the pain.

Evaluation of the Data: The data obtained from the study are SPSS v.22 (Statistical Package for Social Sciences) package program will be used. When parametric test assumptions are fulfilled, repeated measures variance analysis will be used in the analysis of more than two measurements from a group, and Friedman test will be used when parametric test assumptions are not fulfilled. The level of error will be considered as 0.05.

ELIGIBILITY:
Inclusion Criteria:Conscious Open communicable having an tracheal tube or tracheostomy Not using pain medication Patients who do not have a neurological disease that will prevent pain will be included in the study.

-

Exclusion Criteria:Unconscious, communicated but unable to express their pain numerically Using pain medication Patients with neurological diseases that prevent them from feeling pain will not be included in the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
DAS Scor | 30 days
  Whether patients feel pain before and after endotracheal aspiration is evaluated by looking at the patient's movements according to the scale developed by Payen. 3 points express no pain, 12 points express unbearable pain

SECONDARY OUTCOMES:
VAS scor | 90 days
  Whether the patients feel pain before and after the endotracheal aspiration procedure, the patient expresses 0 no pain, 10 unbearable pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gulsoy Z, Ozdemir Kol I. The Effect of Endotracheal Suctioning on Pain in Conscious Adult Patients in Intensive Care Unit. Dimens Crit Care Nurs. 2024 Mar-Apr 01;43(2):72-79. doi: 10.1097/DCC.0000000000000624. PMID 38271311